CLINICAL TRIAL: NCT06508749
Title: Phase I/II Trial to Evaluate the Impact of Three Broadly Neutralizing Antibodies or Analytic Treatment Interruption on Viral Reservoir, Immune Function, and Maintenance of HIV Suppression in Early Treated Children in Botswana
Brief Title: The Tatelo Plus Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2042
Record Dates: First submitted 2024-06-26; First posted 2024-07-18 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: HIV; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1-Step 1a Entry (Experimental): Receiving PGDM1400LS first
  Step 1a includes a single-agent safety lead-in period for PGDM1400LS (Group 1), followed by three bNAbs administered on a rotating schedule while participants continue to receive ART. A pharmacokinetic assessment will be conducted for the three bNAbs.
  Interventions: Drug: PGDM1400LS; Drug: VRC07-523LS; Drug: PGT121.414.LS; Drug: ART Regimen prior to enrolling in Step 1a
- Group 2-Step 1a Entry (Experimental): Receiving PGT121.414.LS first
  Step 1a includes a single-agent safety lead-in period for PGT121.414.LS (Group 2), followed by three bNAbs administered on a rotating schedule while participants continue to receive ART. A pharmacokinetic assessment will be conducted for the three bNAbs.
  Interventions: Drug: PGDM1400LS; Drug: VRC07-523LS; Drug: PGT121.414.LS; Drug: ART Regimen prior to enrolling in Step 1a
- Step 1b Entry (Experimental): ATI Only. For anyone directly enrolling in the Step 3 ATI and not participating in Steps 1 or 2
  In Step 1b participants receive three bNAbs administered on a rotating schedule while continuing to receive ART.
  Interventions: Drug: PGDM1400LS; Drug: VRC07-523LS; Drug: PGT121.414.LS; Drug: ART Regimen prior to enrolling in Step 1b
- Step 2a (Experimental): In Step 2a participants discontinue ART and receive three bNAbs administered on a rotating schedule.
  Interventions: Drug: PGDM1400LS; Drug: VRC07-523LS; Drug: PGT121.414.LS
- Step 2b (Experimental): In Step 2b participants remain off ART and continue to receive three bNAbs administered on a rotating schedule.
  Interventions: Drug: PGDM1400LS; Drug: VRC07-523LS; Drug: PGT121.414.LS
- Step 3 progression (Experimental): ATI Only. Participants discontinue ART and bNAbs. For participants progressing to Step 3 after participating in Steps 1 and 2
  Interventions: Other: Analytic Treatment Interruption
- Group 3- Step 3 Direct Entry (Experimental): ATI Only. Participants discontinue ART. For anyone directly enrolling in the Step 3 ATI and not participating in Steps 1 or 2
  Interventions: Other: Analytic Treatment Interruption

INTERVENTIONS:
Drug: PGDM1400LS — IV Antibody Infusion based on subject's weight
  Arms: Group 1-Step 1a Entry; Group 2-Step 1a Entry; Step 1b Entry; Step 2a; Step 2b
Drug: VRC07-523LS — IV Antibody Infusion based on subject's weight
  Arms: Group 1-Step 1a Entry; Group 2-Step 1a Entry; Step 1b Entry; Step 2a; Step 2b
Drug: PGT121.414.LS — IV Antibody Infusion based on subject's weight
  Arms: Group 1-Step 1a Entry; Group 2-Step 1a Entry; Step 1b Entry; Step 2a; Step 2b
Drug: ART Regimen prior to enrolling in Step 1a — Antiviral drugs are not study product. However, participants will continue to receive the ART regimen they were receiving prior to enrolling in the study during Step 1a.
  Arms: Group 1-Step 1a Entry; Group 2-Step 1a Entry
Drug: ART Regimen prior to enrolling in Step 1b — Antiviral drugs are not study product. However, participants will continue to receive the ART regimen they were receiving prior to enrolling in the study during Step 1b.
  Arms: Step 1b Entry
Other: Analytic Treatment Interruption — (all anti-HIV agents are discontinued)
  Arms: Group 3- Step 3 Direct Entry; Step 3 progression

SUMMARY:
The purpose of this study is to advance pediatric HIV treatment and cure research by evaluating the impact of a combination of three anti-HIV-1 broadly neutralizing antibodies (bNAbs) or analytic treatment interruption (ATI) on viral reservoir, immune function, and maintenance of HIV suppression in early-treated children.

ELIGIBILITY:
Inclusion Criteria, Step 1

* Previously enrolled in the EIT/Tatelo, or Moso Cohort Study
* Receiving prescribed ART for at least 24 weeks prior to study entry as determined by the site investigator based on participant/parent/guardian report and available medical records
* 24 weeks to 12 years of age at enrollment, inclusive
* If entering Step 1a: HIV-1 RNA <40 copies/mL for at least 24 weeks prior to entry, including documented suppression to <40 copies/mL within 30 days of Step 1 entry
* If entering Step 1b: HIV-1 RNA <200 copies/mL for at least 24 weeks prior to entry, including documented suppression to <40 copies/mL within 30 days of Step 1 entry.
* Normal temperature (<37.4°C axillary, or <38°C non-axillary) and no signs or symptoms of acute illness at entry as determined by the site investigator based on participant/parent/guardian report and available medical records
* Normal, grade 1 or grade 2 results for all of the following laboratory tests at screening, based on testing of specimens collected within 30 days prior to entry and grading per protocol:

  * Hemoglobin
  * Absolute neutrophil count
  * Platelet count
  * Alanine aminotransferase
  * Aspartate aminotransferase
  * Creatinine
* For female participants who are able to become pregnant (defined as having reached menarche and not having undergone surgical sterilization), not pregnant based on testing performed from a specimen collected within 5 days prior to enrollment). Note: Pregnancy is not expected in Step 1 given the age range of eligible participants.
* Expected to be available for the duration of participation and expected to comply with the visit schedule and other requirements as determined by the site investigator based on participant/parent/guardian report at entry
* Not currently participating in another study of an investigational agent and is not expected to participate in any such study for the duration of participation, as determined by the site investigator based on participant/parent/guardian report at entry. Prior or current participation in the EIT/Tatelo or Moso cohort studies is permitted.
* Parental/legal guardian is willing and able to provide written permission for child's participation and, child is willing and able to provide written assent for participation if 7- 17 years of age

Inclusion Criteria, Step 2

* At or beyond the Week 24 visit in Step 1
* Susceptible to at least 2 of the 3 bNAbs under study at or prior to Step 1 entry OR Negative EIA and negative qualitative DNA result at last available evaluation in Step 1 in the absence of available susceptibility data
* No confirmed HIV-1 RNA ≥40 copies/mL throughout Step 1 and for at least 24 weeks prior to Step 1 entry

Inclusion Criteria, Step 3

* If entering from Step 1:

  1. At or beyond the Week 24 visit in Step 1, with no confirmed HIV-1 RNA ≥40 copies/mL throughout Step 1
  2. Not eligible for Step 2
  3. No confirmed HIV-1 RNA ≥40 copies/mL for at least 96 weeks prior to Step 3 entry (or since 24 weeks of age if 96-120 weeks of age)
  4. Detection of >80% of intact proviruses in heterochromatin DNA regions (i.e. non-genic DNA, satellite DNA, ZNF genes) from any PBMC sample analyzed by MIP-seq, and no recorded viremia (>40 copies/mL) after this evaluation OR Negative EIA and negative Qualitative HIV DNA result within 12 weeks prior to Step 3 entry
  5. Approved for entry by Clinical Management Committee (CMC)
  6. Willingness and ability to provide independent written informed consent for participation or parental/legal guardian is willing and able to provide written permission for child's participation and, child is willing and able to provide written assent for participation if 7-17 years of age
* If entering from Step 2:

  1. At or beyond the Week 24 visit of Step 2, with HIV-1 RNA <40 copies/mL throughout Steps 1 and 2
  2. No confirmed HIV-1 RNA ≥40 copies/mL for at least 96 weeks prior to Step 3 entry (or since 24 weeks of age if 96-120 weeks of age)
  3. Negative EIA and negative qualitative DNA result within 12 weeks prior to Step 3 entry OR Detection of >80% of intact proviruses in heterochromatin DNA regions (i.e. non-genic DNA, satellite DNA, ZNF genes) from any PBMC sample analyzed by MIP-seq, and no recorded viremia (>40 copies/mL) after this evaluation entry AND approved for entry by CMC
  4. For Moso participants, not currently being breastfed
  5. Willingness and ability to provide independent written informed consent for participation or parental/legal guardian is willing and able to provide written permission for child's participation and, child is willing and able to provide written assent for participation if 7-17 years of age
* If entering Step 3 directly upon enrollment:

  1. Previously enrolled in the EIT/Tatelo, Moso, or BHP Adolescent Cohort Study
  2. 96 weeks to 25 years of age at enrollment, inclusive
  3. "Non-encoding" virus: Detection of >80% of intact proviruses in heterochromatin DNA regions (i.e. non-genic DNA, satellite DNA, ZNF genes) from any PBMC sample analyzed by MIP-seq, and no recorded viremia (>40 copies/mL) after this evaluation OR "No intact virus": adolescent (13-25 years) with no intact HIV detected in at least 20 million PBMCs sampled within the prior 4 years
  4. For "non-encoding" virus: Receiving prescribed ART prior to Step 3 entry, with HIV-1 RNA <40 copies/mL for at least 96 weeks prior to entry (or since 24 weeks of age if 96-120 weeks of age), including documented suppression to <40 copies/mL within 30 days of Step 3 entry
  5. For "no intact virus": Receiving prescribed ART prior to Step 3 entry, with HIV-1 RNA <40 copies/mL for at least 10 years prior to entry, including documented suppression to <40 copies/mL within 30 days of Step 3 entry
  6. Approved for entry by CMC
  7. For Moso participants, not currently being breastfed
  8. For female participants who are able to become pregnant (defined as having experienced menarche and not having undergone surgical sterilization), not pregnant based on testing performed from a specimen collected within 5 days prior to enrollment)
  9. For female participants who are able to become pregnant (defined as having reached menarche and not having undergone surgical sterilization) and report sexual activity that could lead to pregnancy, willing to use two methods of contraception while on study. One of the two methods must be highly effective; highly effective methods include the following:

     * Contraceptive intrauterine device or intrauterine system
     * Subdermal contraceptive implant
     * Progestogen injections
     * Combined estrogen and progestogen oral contraceptive pills
     * Percutaneous contraceptive patch
     * Contraceptive vaginal ring The highly effective method must be initiated prior to enrollment. The second method must be a barrier method for dual protection against pregnancy and to avoid transmission of HIV during the ATI and other sexually transmitted infections.
  10. For female participants who are able to become pregnant, not currently breastfeeding an infant, and not intending to breastfeed an infant for the duration of the study, based on participant/parent/guardian report at entry
  11. For participants who report sexual activity, willing to receive counseling and to use condoms to avoid transmission of HIV
  12. Expected to be available for the duration of participation and expected to comply with the visit schedule and other requirements as determined by the site investigator based on participant/parent/guardian report at entry
  13. Not currently participating in another study of an investigational agent and is not expected to participate in any such study for the duration of participation, as determined by the site investigator based on participant/parent/guardian report at entry. Prior or current participation in the EIT/Tatelo, Moso, or BHP Adolescent cohort studies is permitted.
  14. Willingness and ability to provide independent written informed consent for participation or parental/legal guardian is willing and able to provide written permission for child's participation and, child is willing and able to provide written assent for participation if 7-17 years of age

Inclusion Criteria, Step 4

* Previously entered the study in Step 1 or Step 3. All participants will enter Step 4 upon completing a prior study step. Participants ending Step 1a or Step 1b who, for any reason, do not proceed to Step 2 or to Step 3 will be eligible to proceed to Step 4. Participants ending Step 2 who, for any reason, do not proceed to Step 3 will be eligible to proceed to Step 4. Participants ending Step 3 for any reason will be eligible to proceed to Step 4.

Exclusion Criteria:

* Active tuberculosis (either suspected or proven) or malignancy.
* Hepatitis B surface antigen (HBsAg) positive
* Received within 30 days prior to study entry, or is identified as requiring, any of the following:

  * Any immunoglobulin-based treatment
  * Chronic (more than 14 days) systemic steroid treatment
* Has any other documented or suspected clinically significant medical condition or any other condition that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* For participants entering Step 1 and Step 2: <5 kg or >115kg.
* For participants entering Step 3 directly: Received NNRTI-based ART (including efavirenz, nevirapine, rilpivirine) within 14 days of Step 3 entry

Ages: 24 Weeks to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-11-05 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
To describe the safety and pharmacokinetics of bNAb immunotherapy with VRC07-523LS, PGDM1400LS and PGT121.414.LS when added to existing effective ART in early-treated children living with HIV-1 in Botswana | Through week 32
  Occurrence of Grade 3 or higher adverse events Occurrence of Grade 1 or higher bNAb-related adverse events Occurrence of any SAE Permanent discontinuation of study product Pre-dose trough concentrations of VRC07-523LS, PGDM1400LS and PGT121.414.LS at Week 16 Pre-dose trough concentrations of VRC07-523LS, PGDM1400LS and PGT121.414.LS through 32 weeks
To describe the safety of up to 24 weeks of bNAb immunotherapy with VRC07-523LS, PGDM1400LS and PGT121.414.LS when added on a rotating schedule to existing effective ART in early-treated children living with HIV-1 in Botswana | Through week 24
  Occurrence of Grade 3 or higher adverse events Occurrence of Grade 1 or higher bNAb-related adverse events Occurrence of any SAE Permanent discontinuation of study product
To determine the safety of 24 weeks of maintenance VRC07-523LS, PGDM1400LS and PGT121.414.LS immunotherapy alone, following the discontinuation of ART | Through Week 24
  Occurrence of Grade 3 or higher adverse events Occurrence of Grade 1 or higher bNAb-related adverse events
To determine the maintenance of virologic suppression of 24 weeks of maintenance VRC07-523LS, PGDM1400LS and PGT121.414.LS immunotherapy alone, following the discontinuation of ART | Through Week 24
  Viral rebound defined as plasma HIV-1 RNA ≥400 copies/mL at or prior to 24 weeks of bNAb-only treatment.
To determine the CD4 cell count preservation of 24 weeks of maintenance VRC07-523LS, PGDM1400LS and PGT121.414.LS immunotherapy alone, following the discontinuation of ART | Through Week 24
  Change in absolute CD4 cell count
To describe the safety, maintenance of virologic suppression, and CD4 cell count preservation of up to 48 weeks of ATI (with no ART or bNAbs) among participants who meet specified criteria for an ATI | Through Week 48
  Occurrence of Grade 3 or higher adverse events Occurrence of Grade 1 or higher ATI-related adverse events Viral rebound defined as plasma HIV-1 RNA ≥400 copies/mL at or prior to 48 weeks of ATI Change in absolute CD4 cell count

SECONDARY OUTCOMES:
To measure the proportion of participants with viral rebound defined as a single plasma HIV-1 RNA ≥400 copies/mL at or prior to 48 weeks of bNAb-only treatment (for those who continue bNAb-only treatment beyond 24 weeks) | Through week 48
  Viral rebound defined as plasma HIV-1 RNA ≥400 copies/mL at or prior to 48 weeks of bNAb-only treatment (among participants who continue beyond 24 weeks on bNAb-only treatment)
To monitor and report time to re-suppression of plasma HIV-1 RNA following re-initiation of ART, for participants who experience viral rebound on bNAbs alone or during ATI | Through week 48
  Time to viral re-suppression defined as first HIV-1 RNA <40 copies/mL following ART resumption
To measure the size of residual viral reservoirs, during each step of the study. Comparisons will include change during triple bNAbs + ART; change during triple bNAbs alone; change during ATI; and change during entire study | Through week 48
  Change in total, intact, and defective provirus between entry and end of triple bNAbs + ART Change in total, intact, and defective provirus between start of bNAb-only treatment and end of bNAb-only treatment Change in total, intact, and defective provirus between start of ATI and end of ATI.
  Change in total, intact, and defective provirus between study entry and end of ATI.

CONTACTS AND LOCATIONS:
Locations (2):
- Botswana (2):
  - Francistown CRS (CRS #31891), Francistown
  - Botswana Harvard Health Partnership CRS (CRS #31833), Gaborone

IPD SHARING:
Plan to Share IPD: Yes
individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: Researchers who provide a methodologically sound proposal for use of the data that is approved by the protocol leadership.
  * For what types of analyses?
  * To achieve aims in the proposal approved by the protocol leadership.
  * By what mechanism will data be made available?
  * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https:// www.impaactnetwork.org/ resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.